CLINICAL TRIAL: NCT02995863
Title: Clinical Efficacy of Therapeutic Footwear With a Rigid Rocker Sole in the Prevention of Reulceration in Patients With Diabetes Mellitus and Diabetic Polineuropathy: a Prospective and Randomized Clinical Trial.
Brief Title: This Research Hypothesizes That the Use of a Rigid Rocker Sole Reduces the Recurrence Rate of Diabetic Foot Ulcers in Patients With Peripheral Neuropathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Mateo López Moral, Clinical Research, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UComplutenseMadrid
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

ARMS (2):
- Experimental Group (Experimental): Rigid rocker sole footwear
  Interventions: Device: Rigid Rocker Sole Footwear
- Control Group (Active Comparator): Therapeutic footwear
  Interventions: Device: Therapeutic Footwear

INTERVENTIONS:
Device: Rigid Rocker Sole Footwear
  Arms: Experimental Group
Device: Therapeutic Footwear
  Arms: Control Group

SUMMARY:
This research presents a randomized clinical trial which analyzes the efficacy of a rigid rocker sole in the reduction of the recurrence rate of plantar ulcers in diabetic foot patients. The hypothesis of the research is the use of a rigid rocker sole reduces the recurrence rate of diabetic foot ulcers in patients with peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetic patients regardless of the pharmacotherapy that they receive.
* Adult patients of both sexes.
* Peripheral neuropathy patients.
* Patients without wounds or ulcers at the examination time.
* Patients with a foot ulcers history.
* Patients with or without minor amputation prior to the inclusion time in the present study.
* Patients who don´t need gait support mechanisms such as walking sticks, crutches, splints or any other devices which interferes with the autonomous development of the gait.

Exclusion Criteria:

* Patients with mayor amputation.
* Patients with rheumatic disease that affect the feet.
* Patients with peripheral neuropathy of different etiology to Diabetes mellitus.
* Patients with several critical ischemia criteria, defined by TACS II guideline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Presence of diabetic foot ulcer | through study completion, an average of 6 months
  The Wagner system assesses ulcer depth and the presence of osteomyelitis or gangrene using the following grades: grade 0 (pre- or post-ulcerative lesion), grade 1 (partial/full-thickness ulcer), grade 2 (probing to tendon or capsule), grade 3 (deep with osteitis), grade 4 (partial foot gangrene) and grade 5 (whole foot gangrene

SECONDARY OUTCOMES:
Ankle Joint movility | through study completion, an average of 6 months
  The ankle joint is examined in the neutral position, with the patient prone; a vertical line is marked on the patient's skin from heel to midcalf, and the maxi- mum range of dorsiflexion in passive motion is mea- sured in degrees with a goniometer. The normal value for the ankle joint is a mobility >90° of dorsi- flexion.
Mobility of the First metatarsal Joint | through study completion, an average of 6 months
  Is examined with the patient in the supine position, and a horizontal line is drawn from the big toe to the heel. The maximum range of pas- sive dorsiflexion is recorded. The normal range of joint mobility is >65° at rest and 30° when the patient is standing.
Subtalar Joint Movements | through study completion, an average of 6 months
  (inversion and eversion) are examined with the patient in a prone position, holding the calcaneus with one hand and the neck of the astragalus with the thumb and index finger of the other hand. Holding the astragalus rather than the tibia isolated the s
IPAQ (International Physical Activity Questionnaires) | through study completion, an average of 6 months
  The purpose of the International Physical Activity Questionnaires (IPAQ) is to provide a set of well-developed instruments that can be used internationally to obtain comparable estimates of physical activity. There are two versions of the questionnaire. The short version is suitable for use in national and regional surveillance systems and the long version provide more detailed information often required in research work or for evaluation purposes.
Foot Type | through study completion, an average of 6 months
  The validated protocol of the Foot Posture Index-6 involves the rating of three criteria in the rearfoot: Talar head palpation,Supra- and infra-lateral malleolar curvature and Calcaneal frontal plane position. In addition, there are three criteria on the forefoot: Prominence in the region of the talonavicular joint (TNJ), Congruence of the medial longitudinal arch (MLA), Abduction/adduction of the forefoot on the rearfoot. Each item is graded by a five-point Likert-type, from -2 to +2: 0 for neutral, with a minimum score of -2 for clear signs of supination, and +2 for positive signs of pronation. The final FPI-6 score will be a whole number between -12 and +12. A total FPI-6 score between 0 and +5 indicates a neutral foot, a score of above +6 indicates a pronated or highly pronated foot, and a score between -1 and -12 indicates a supinated or highly supinated foot.
Deformities | through study completion, an average of 6 months
  Forefoot deformities were considered when the foot presented any of the following: hallux valgus, Tailor's bunion; toe contractures (hammer-toe, claw-toe or mallet-toe deformities); subluxation or dislocation of the metatarsophalangeal joints (overlapped toe and prominent metatarsal heads).
Ankle - Brachial Index (ABI) | through study completion, an average of 6 months
  Were assessed by the same experienced podiatrist using a manual 8 MHz Doppler (Doppler II, Huntleigh Healthcare Ltd, South Glamorgan, UK), and the toe systolic pressure was taken with a digital plethysmography (Systoe, Atys Medical, Quermed, Madrid). The dorsalis pedis artery was used for recording ankle values. The ABI were calculated with the equations of the ankle pressure readings divided by the highest brachial reading between the right and left arms. We considered Peripheral Arterial Disease to have an ABI value less than 0.9; normal ABI values were between 0.9 and 1.39, and an ABI value ≥1.4 was considered poorly compressible vessels related to medial arterial calcification in distal arteries.
Sensorimotor neuropathy | through study completion, an average of 6 months
  Sensorimotor neuropathy was diagnosed by evaluation using a Semmes-Weinstein 5.07/10 g monofilament and a biothesiometer (both from Novalab Iberica, Madrid, Spain). Patients who did not feel 1 of the 2 tests were diagnosed with neuropathy.
Physical Activity Questionnaire | through study completion, an average of 6 months
  Measurements about time of use of footwear either at home or outdoor. Normal value ranges are: never, 1 day per week, 1 to 3 day per week, 4 to 5 days per week and 6 to 7 days per week.
  And measurements about how many hours per day the patient wear the footwear, the normal value ranges are: less than 1 hour, 1 to 3 hours per day, 4 to 7 hours per day, 8 to 11 hours per day and more than 12 hours per day.
Toe - Brachial Index (TBI) | through study completion, an average of 6 months
  Were assessed by the same experienced podiatrist using a manual 8 MHz Doppler (Doppler II, Huntleigh Healthcare Ltd, South Glamorgan, UK), and the toe systolic pressure was taken with a digital plethysmography (Systoe, Atys Medical, Quermed, Madrid). The ABI and the TBI were calculated with the equations of the ankle or toe pressure readings divided by the highest brachial reading between the right and left arms. We considered PAD to have a TBI value less than 0.7; normal TBI values were between 0.7 and 0.99, and TBI ≥ 1 was considered distal arteries calcification.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitaria de Podología de la Universidad Complutense de Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lopez-Moral M, Lazaro-Martinez JL, Garcia-Morales E, Garcia-Alvarez Y, Alvaro-Afonso FJ, Molines-Barroso RJ. Clinical efficacy of therapeutic footwear with a rigid rocker sole in the prevention of recurrence in patients with diabetes mellitus and diabetic polineuropathy: A randomized clinical trial. PLoS One. 2019 Jul 11;14(7):e0219537. doi: 10.1371/journal.pone.0219537. eCollection 2019. PMID 31295292